CLINICAL TRIAL: NCT02189447
Title: Photorefractive Keratectomy and Corneal Cross-linking in Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEC 126
Record Dates: First submitted 2014-07-05; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Keratoconus
Keywords: Keratoconus; Ectasia; Corneal Cross-linking
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refractive surgery (Experimental): Patients with keratoconus treated with simultaneous photorefractive keratectomy and Corneal collagen cross-linking.
  Interventions: Procedure: Simultaneous Photorefractive Keratectomy and Collagen Cross-linking in patients with keratoconus

INTERVENTIONS:
Procedure: Simultaneous Photorefractive Keratectomy and Collagen Cross-linking in patients with keratoconus — Photorefractive Keratectomy followed by Collagen Cross-linking in patients with keratoconus in the same surgical setting

SUMMARY:
Evaluation of the safety and efficacy of surface ablation followed by Collagen Cross-linking in patients with keratoconus

ELIGIBILITY:
Inclusion Criteria:

* contact lens intolerance
* corneal thickness > 450 micrometers
* Keratometry < 56 diopters
* Astigmatism < 6 diopters

Exclusion Criteria:

* corneal thickness < 450 micrometers
* Keratometry > 56 diopters
* Astigmatism > 6 diopters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The change of visual acuity following Photorefractive Keratectomy and Corneal Collagen Cross-linking in patients with Keratoconus | 6 months
  The change of visual acuity from baseline in patients suffering from keratoconus following treatment with Photorefractive Keratectomy and Corneal Collagen Cross-linking.